CLINICAL TRIAL: NCT06298734
Title: Modulating Immune-Microbiome Axis Through High-Intensity Exercise and High-Fiber Diet for Immunotherapy Outcomes in Melanoma Patients: The DUO Trial
Brief Title: High-Intensity Exercise and High-Fiber Diet for Immunotherapy Outcomes in Melanoma Patients: The DUO Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: World Cancer Research Fund International (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-712
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Melanoma (Skin); Skin Cancer; Advanced Melanoma
Keywords: Melanoma; Skin Cancer; Advanced Melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: High-Intensity Exercise (EX) (Experimental): 10 participants will complete:
  * In-office baseline visit.
  * Virtual exercise sessions 3x weekly.
  * Post-intervention in-office visit.
  Interventions: Behavioral: Exercise Program
- Group B: High-Fiber Diet (DT) (Experimental): 10 participants will complete:
  * In-office baseline visit.
  * 1x weekly appointment with research staff to review to review diet adherence.
  * Post-intervention in-office visit.
  Interventions: Behavioral: Diet Program
- Group C: Combined High-Intensity Exercise and High-fiber Diet (COMB) (Experimental): 10 participants will complete:
  * In-office baseline visit.
  * Virtual exercise sessions 3x weekly.
  * 1x weekly appointment with research staff via Zoom platform to review to review diet adherence. Diet appointment may be combined with exercise session appointment.
  * Post-intervention in-office visit.
  Interventions: Behavioral: Exercise Program; Behavioral: Diet Program
- Group D: Attention Control (AC) (No Intervention): 10 participants will complete:
  * In-office baseline visit.
  * Participants will receive a general healthy lifestyle guidebook.
  * Pot-intervention in-office visit.

INTERVENTIONS:
Behavioral: Exercise Program — A high-intensity interval training, aerobic exercise program virtually supervised, home-based, and appointment-based program under direct one-on-one supervision by a trained oncology exercise specialist. Sessions will be conducted via the Zoom platform. Participants will be provided with home stationary bike, heart rate monitor, blood pressure monitor. For participants who do not have a smart device, a Wi-Fi enabled tablet will be provided.
  Arms: Group A: High-Intensity Exercise (EX); Group C: Combined High-Intensity Exercise and High-fiber Diet (COMB)
Behavioral: Diet Program — A virtual dietary consultation program supervised by trained research staff. Appointments will be conducted via the Zoom platform. Participants will receive an education handout at the baseline visit.
  Arms: Group B: High-Fiber Diet (DT); Group C: Combined High-Intensity Exercise and High-fiber Diet (COMB)

SUMMARY:
The purpose of this study is to determine whether high-intensity exercise and high-fiber diet are feasible and improve various health outcomes among participants with advanced melanoma receiving immunotherapy.

The names of the groups in this research study are:

* High-Intensity Exercise (EX)
* High-fiber Diet (DT)
* Combined High-Intensity Exercise and High-Fiber Diet (COMB)
* Attention Control (AC)

DETAILED DESCRIPTION:
This single-center, four-arm, pilot randomized research study is to test if high-intensity exercise and high-fiber diet are feasible and effective in improving the gut microbiome health, immune function, physical fitness, treatment-related side effects, and treatment outcomes in participants with advanced melanoma receiving immunotherapy. Participants will be randomized into 1 of 4 study groups: Group A Exercise, Group B Diet, Group C Combined, and Group D Attention Control. Randomization means a participant will be placed into an intervention group by chance.

The information learned by doing this research may help determine whether participating in such lifestyle interventions are tolerable during immunotherapy and exert health benefits among melanoma participants.

The research study procedures include screening for eligibility, study visits, stool samples, blood tests, and questionnaires.

Participation in this study is expected to last up to a total of 9 weeks.

It is expected about 40 people will take part in this research study.

This study is sponsored by the World Cancer Research Fund International.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; due to the rarity of the disease in those <18 years, this age bracket will not be included.
* Histologically diagnosed with advanced melanoma.
* Having been or newly receiving immune checkpoint inhibitor, including anti-PD1, antiCTLA4, and/or anti-LAG3 monoclonal antibodies, with palliative intent for at least one month with a plan to continue immunotherapy for at least 8 weeks (i.e., study intervention period) at the time of recruitment.
* Not receiving other concurrent tumor-directed systemic treatment (e.g., chemotherapy or targeted therapy).
* Medically cleared to participate in high-intensity exercise and high-fiber diet by their treating oncologist.
* Not having medical conditions that could exacerbate with exercise, such as bone disease at imminent risk of fracture or uncontrolled cardiopulmonary or metabolic diseases (e.g., uncontrolled hypertension or diabetes).
* Currently not meeting the physical activity guideline (i.e., more than 150 minutes per week of moderate-to-vigorous intensity, regular, structured aerobic exercise) over the past month at the time of recruitment.
* Currently not meeting the daily dietary fiber intake guideline (i.e., 30 grams/day) over the past month at the time of recruitment.
* Ability to communicate and complete written forms in English.
* Ability to understand and the willingness to sign informed consent prior to any study- related procedures.
* Willing to travel to DFCI for necessary data collection.

Exclusion Criteria:

* Receiving other concurrent systemic treatment for advanced melanoma such as chemotherapy or targeted therapy. This study is to exclusively target patients receiving immune checkpoint inhibitors where other treatments may impact the study outcomes of intervention efficacies and feasibilities.
* Participating in more than 150 minutes of moderate-to-vigorous aerobic exercise per week over the past month. This study targets insufficiently active persons to assess the effect of the described exercise intervention, where additional exercise done regularly will contaminate the intervention outcomes.
* Consuming more than 25 and 38 grams of dietary fiber per day for women and men, respectively over the past month. This study targets persons who insufficiently take dietary fiber to assess the effect of the described dietary intervention, where additional dietary fiber intake will contaminate the intervention outcomes.
* Having unstable comorbidities or medical conditions that prevent participation in high intensity exercise or high-fiber diet interventions. Patients with unstable medical conditions may develop unexpected adverse events from exercise and dietary changes. For the purpose of patients' safety, patients with unstable medical conditions are excluded.
* Subjects who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
* Development of second malignancy (except for basal cell carcinoma or squamous cell carcinoma of the skin) that requires concurrent treatment, which would interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Gut Microbiome Diversity | Baseline (Week 1) and post-intervention (Week 10)
  The primary outcome of the study is the gut microbiome diversity measured by the Shannon Diversity Index. Alpha diversity of samples will be quantified using the Shannon diversity index, and beta diversity will be quantified using the Bray-Curtis dissimilarity.

SECONDARY OUTCOMES:
Change in Systemic Immune Function | Baseline (Week 1) and post-intervention (Week 10)
  Immune phenotyping will be conducted using the blood samples drawn at baseline and post-intervention. Immunofluorescence will be performed using a flow cytometry, which analyzes the physical and fluorescent properties of cells in suspension in real-time as they flow through the instrument.
Change in Cardiopulmonary Fitness | Baseline (Week 1) and post-intervention (Week 10)
  Cardiorespiratory fitness will be assessed as VO2peak by a graded maximal cycle exercise stress test. VO2peak is defined as the highest values of oxygen uptake averaged among every 15-second interval during the test.
Change in Short Physical Performance Battery (SPPB) | Baseline (Week 1) and post-intervention (Week 10)
  Physical function will be assessed by the SPPB. This includes the following 3 lower extremity measures completed in the following order. Timed balance (seconds): Balance will be assessed under 3 conditions (side-by-side, semi-tandem, and tandem stands). Gait speed (seconds): Gait speed will be assessed over a 4-meter flat surface distance. The participant will be asked to complete 2 attempts of this test. Time will be recorded using an electronic timing system. Chair stand (seconds): Chair stand will be performed under 2 conditions: a) subjects will perform a single chair stand; b) subjects will be asked to perform 5 repeated chair stands as quickly as possible; time to completion will be recorded.
Change in Percent Body Fat | Baseline (Week 1) and post-intervention (Week 10)
  Percent body fat will be assessed via bioelectrical impedance using a validated device (Tanita 780, Arlington Heights, IL). Participants will be asked to remove their shoes and socks and stand still on the device while holding the handles with their hands at their sides. The device will estimate body fat using an algorithm based on age, sex, height, and body weight.
Change in Lean mass | Baseline (Week 1) and post-intervention (Week 10)
  Lean mass (kg) will be assessed via bioelectrical impedance using a validated device (Tanita 780, Arlington Heights, IL). Participants will be asked to remove their shoes and socks and stand still on the device while holding the handles with their hands at their sides. The device will estimate body fat using an algorithm based on age, sex, height, and body weight.
Change in Hip circumference | Baseline (Week 1) and post-intervention (Week 10)
  A constant-tension tape measure will be used to obtain waist circumference (i.e., the distance around the waist using the umbilicus as the reference point) (cm).
Change in Waist circumference | Baseline (Week 1) and post-intervention (Week 10)
  A constant-tension tape measure will be used to obtain hip circumference (the distance around the widest girth of the buttocks using the greater trochanter as a landmark) (cm).
Change in Health-Related Quality of life (EORTC-QLQ C30) | Baseline (Week 1) and post-intervention (Week 10)
  The European Organization for Research and Treatment of Cancer- Quality of Life Questionnaire-C30 will assess health-related quality of life, consisting of subscales including functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures. The score ranges from 0 to 100 and a higher value indicates a better quality of life.
Change in MDASI-Immunotherapy Questionnaire Score | Baseline (Week 1) and post-intervention (Week 10)
  MD Anderson Symptom Inventory-Immunotherapy (MDASI-Immunotherapy EPT) module is comprised of 20 symptoms including 7 immunotherapy-specific items in addition to the 13 MDASI core symptoms.The MDASI asks participants to rate the severity of disease-related and treatment-related symptoms during the past 24 h. Each symptom (pain, fatigue, nausea, disturbed sleep, emotional distress, shortness of breath, difficulty remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, numbness or tingling, rash, diarrhea, pain the abdomen, swelling in the hands and legs, headache, night sweats and fever and/or chills) is rated on an 11-point scale ranging from 0 (not present) to 10 (as bad as you can imagine). The MDASI-Immunotherapy EPT has been shown to be valid and reliable.
Change in Anxiety (HADS) | Baseline (Week 1) and post-intervention (Week 10)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-question instrument that measures anxiety and depression with seven questions for each. Each question is scored between zero (no impairment) and three (severe impairment), with a maximum score of 21 for anxiety.
Change in Depression (HADS) | Baseline (Week 1) and post-intervention (Week 10)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-question instrument that measures anxiety and depression with seven questions for each. Each question is scored between zero (no impairment) and three (severe impairment), with a maximum score of 21 for depression.
Change in Sleep Quality (PSQI) | Baseline (Week 1) and post-intervention (Week 10)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The PSQI contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. The seven components are then summed to obtain a global score ranging from 0-21 points.
Proportion of Participants Completing the Exercise Intervention Sessions | Post-intervention (Week 10)
  The primary outcome is feasibility and will be assessed by the proportion of participants completing the exercise intervention sessions with >70% completion considered feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu